CLINICAL TRIAL: NCT07021859
Title: Induction of Migraine Attacks With Aura Using Calcitonin Gene-Related Peptide: A Randomized Clinical Trial
Brief Title: Induction of Migraine Attacks With Aura Using Calcitonin Gene-Related Peptide
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Haidar Al-Khazali, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-23042433
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Migraine Aura; Migraine With Aura
Keywords: Migraine; Aura; Calcitonin gene-related peptide
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders; Epilepsy | interventions — Calcitonin

STUDY DESIGN:
Intervention Model Description: This single-center trial applies a randomized, double-blind, placebo-controlled, two-way crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcitonin gene-related peptide (CGRP) (Experimental): CGRP will be administered by intravenous infusion.
  Interventions: Drug: Calcitonin-gene related peptide (CGRP)
- Placebo (Placebo Comparator): Placebo (isotonic saline) will be administered by intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitonin-gene related peptide (CGRP) — The participants will receive a continuous intravenous infusion of 1.5 μg/min of CGRP over 60 minutes.
  Arms: Calcitonin gene-related peptide (CGRP)
Drug: Placebo — The participants will receive a continuous intravenous infusion of 60 mL of placebo (isotonic saline) over 60 minutes.
  Arms: Placebo

SUMMARY:
Calcitonin gene-related peptide (CGRP) is a key neuropeptide in migraine pathophysiology and treatment. This study investigates whether CGRP administration can trigger aura in individuals with a diagnosis of migraine with aura.

DETAILED DESCRIPTION:
Recent open-label findings show that calcitonin gene-related peptide (CGRP), a key player in migraine, can trigger aura attacks-despite its limited ability to cross the blood-brain barrier. This suggests CGRP might induce migraine aura via trigeminovascular activation, the same pathway involved in migraine headache. If confirmed, this could reshape treatment strategies for patients diagnosed with migraine with aura. To validate this effect and rule out nocebo influence, a randomized, double-blind, placebo-controlled trial is essential. Its outcomes could inform future therapies targeting the migraine-aura connection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years of age upon entry into screening
* History of migraine with aura for ≥ 12 months according to the International Classification of Headache Disorders 3rd Edition (ICHD-3) criteria
* ≥ 1 monthly day with aura that meets criteria as aura on average across the three months before screening
* Provision of informed consent prior to initiation of any study-specific activities/procedures.

Exclusion Criteria:

* Any history of a primary or secondary headache disorder other than migraine without aura, migraine with aura, chronic migraine, and episodic tension-type headache
* History or evidence of any other clinically significant disorder, condition, or disease (except for those outlined above) that, in the opinion of the site investigator, would pose a risk to subject safety or interfere with study evaluation, procedures or completion
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior
* Female subjects of childbearing potential with a positive pregnancy test during any study visit
* Cardiovascular disease of any kind, including cerebrovascular diseases
* Hypertension (systolic blood pressure of ≥150 mmHg and/or diastolic blood pressure of ≥100 mmHg) prior to the start of infusion on the experimental day
* Hypotension (systolic blood pressure of ≤90 mmHg and/or diastolic blood pressure of ≤50 mmHg)
* Initiation, discontinuation, or change of dosing of prophylactic medications within 2 months prior to study inclusion
* Intake of acute medications (e.g. analgesics, triptans) within 48 hours of infusion start
* Headache of any intensity within 48 hours of infusion start
* Aura within 48 hours of infusion start

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of migraine attacks with aura | 12 hours
  Difference in incidence of migraine attack with aura between CGRP and placebo during the 12-hour observational period after infusion start.

SECONDARY OUTCOMES:
Incidence of migraine attacks without aura | 12 hours
  Difference in incidence of migraine headache between CGRP and placebo during the 12-hour observational period after infusion start.
Headache intensity scores | 12 hours
  Difference in area under the curve (AUC) for headache intensity scores between CGRP and placebo during the 12-hour observational period after infusion start.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data not published within this article will be made available on reasonable request from any qualified investigator.